CLINICAL TRIAL: NCT03746119
Title: Acute Vascular Effects of Short-term E-cigarette Inhalation
Brief Title: Acute Vascular Effects of E-cigarette Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jenny Bosson, MD; PhD, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Umu-2019-31M
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: Nicotine; Electronic cigarette; E-cigarrette; Forearm Plethysmography
MeSH Terms: conditions — Vaping | interventions — E-Cigarette Vapor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine-free e-cigarette (Active Comparator): Subjects will undergo baseline assessments, then actively inhale nicotine-free vapor from an e-cigarette prior to blood samples and various cardiovascular testing.
  Interventions: Other: E-cigarette vapor, nicotine free
- Nicotine e-cigarette (Active Comparator): Subjects will undergo baseline assessments, then actively inhale nicotine containing vapor from an e-cigarette prior to blood samples and various cardiovascular testing.
  Interventions: Other: E-cigarette vapor containing nicotine

INTERVENTIONS:
Other: E-cigarette vapor containing nicotine — A fourth generation e-cigarette device will be used with pre-determined temperature, voltage and wattage settings, and pre-mixed e-solution containing nicotine.
  Arms: Nicotine e-cigarette
Other: E-cigarette vapor, nicotine free — A fourth generation e-cigarette device will be used with pre-determined temperature, voltage and wattage settings, and pre-mixed nicotine free e-solution.
  Arms: Nicotine-free e-cigarette

SUMMARY:
Tobacco use harms nearly every organ in the body and has been linked to ischemic heart disease, chronic obstructive pulmonary disease, stroke, respiratory illness, lung cancer and other cancers. The World Health Organization estimates that 6 million people worldwide lose their lives due to tobacco use yearly, making cigarette smoking one of the leading single causes of preventable death and morbidity.

As this knowledge becomes more common and wide-spread the sales of cigarettes has seen a decrease in recent years. On account of this, the electronic cigarette (e-cigarette) has been introduced to the market as an alternative to traditional cigarette smoking. Electronic cigarettes, also known as e-cigarettes or e-cigs, are delivery devices which heat a base liquid, to which nicotine and flavorings can be added, into vapor which is then inhaled ("vaping"). E-cigarettes have been aggressively marketed as a cheaper, healthier, cleaner alternative to smoking in both advertising and media outlets, primarily targeting adolescents.

Despite growing e-cigarette use, scientific data on health effects are insufficient in some respects and completely lacking in others. However, the investigators have recently shown that cigarette smoking, as well as e-cigarette inhalation, both cause an acute increase of endothelial progenitor cells (EPCs) in the blood of healthy volunteers, suggesting vascular injury, inflammation and a negative impact on hemostasis.

Therefore, using well validated methods, including forearm plethysmography, biomarkers in blood, arterial stiffness measurements and microcirculation assessment (GlycoCheck), the investigators aim to further investigate the effects of e-cigarette inhalation on the vascular system. These measurements will be performed before and after healthy subjects inhale vapor from a e-cigarette on two separate occasions, with and without nicotine in a double-blinded, randomized protocol.

DETAILED DESCRIPTION:
According to the World Health Organization cigarette smoking is today one of the leading single causes of preventable death and morbidity. It is estimated that 7 million people worldwide lose their lives due to tobacco use yearly. On average, cigarette smokers are estimated to die 10 years earlier than non-smokers. Ischemic heart disease, chronic obstructive pulmonary disease, stroke, respiratory illness, lung cancer and other cancers have all been linked to tobacco use. Cigarette smoking has known detrimental effects on the blood vessels and both active as well as passive use causes endothelial dysfunction, one of the earliest signs of atherosclerosis. The investigators have recently shown that cigarette smoking, as well as e-cigarette inhalation, both cause an acute increase of endothelial progenitor cells (EPCs) in the blood of healthy volunteers, suggesting vascular injury, inflammation and negative impact on hemostasis.

In recent years the electronic cigarette has been introduced to the market as an alternative to traditional cigarette smoking. Electronic cigarettes, also known as e-cigarettes or e-cigs, are nicotine delivery devices, which heat a base liquid, to which nicotine and flavorings can be added, into vapor which is then inhaled ("vaping"). Many of the first generation e-cigs emulate conventional cigarettes in appearance, though in second and third generation devices many shapes and sizes exist, varying from one time devices roughly the size of a conventional cigarette to much larger atomizers, designed to be refilled. E-cigarettes have been aggressively marketed as a cheaper, healthier, cleaner alternative to smoking in both advertising and media outlets, primarily targeting women and adolescents.

With declining cigarette sales in the western world, tobacco companies show a great interest in this expanding and highly profitable market, buying already established e-cigarette companies. In February 2014, the European Commission revised the tobacco products directive allowing the trade of e-cigarettes in the European Union. Despite growing e-cigarette use, scientific data on health effects are insufficient in some respects and completely lacking in others. With limited knowledge of e-cigarette vaping health effects in humans it has been challenging for governments and health officials to give advice and regulate the use of this novel product. Therefore, using the 'gold standard' method for assessing vascular function, forearm plethysmography, the investigators aim to investigate the effects of e-cigarette inhalation on the cardiovascular system.

Healthy volunteers will attend on three occasions. The initial visit will be a health assessment in order for inclusion into the study, when ECG, spirometry and blood sampling (max 30 ml of blood) will be performed.

All subjects will inhale vapor from a nicotine-containing e-cigarette for 30 minutes in a specially prepared room with adequate ventilation. In a randomized cross-over fashion, subjects will also 'smoke' e-cigarette without nicotine on separate occasions. These two occasions will be separated by at least one week.

Subjects will rest for 20 minutes prior to vaping. Arterial stiffness, blood pressure, microcirculation assessment (GlycoCheck) and pulse will be measured before and for 60 minutes following vaping. Blood samples will be drawn before, as well as at several time points throughout the study protocol.

Forearm blood flow will be measured using venous occlusion plethysmography in both forearms before and during the intra-arterial infusion of acetylcholine (5, 10 & 20 µg/min; an endothelial-dependent, NO- dependent vasodilator), glyceryl trinitrate (4, 8 & 16 nmol/min; an endothelial-independent, NO-dependent vasodilator), and bradykinin (100, 300 & 1000 pmol/min; an endothelial-dependent vasodilator that stimulates release of tissue plasminogen activator (t-PA)).

ELIGIBILITY:
Inclusion Criteria:

* Intermittent/sporadic use of forms of nicotine
* Normal clinical examination
* Normal EKG
* Normal blood tests
* Normal lung function

Exclusion Criteria:

* Diagnosed cardiovascular disease
* Diagnosed respiratory disease
* Diagnosed systemic or chronic disorders such as rheumatologic or metabolic disease
* Symptoms of infection or inflammation within 2 weeks of the study
* BMI≥30

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Vascular vasomotor function | 3 hours
  Forearm venous occlusion plethysmography to measure forearm blood flow during unilateral intrabrachial infusion of endothelial-dependent and -independent vasodilators. Assessment is shown in ml/100ml tissue/min.

SECONDARY OUTCOMES:
Arterial Stiffness | 1 hour
  Pulse wave analysis (PWA) will be assessed.
Arterial Stiffness | 1 hour
  Pulse wave velocity (PWV) will be assessed.
Cotinine Cardiovascular biomarkers Cardiovascular biomarkers | 6 hours
  Blood samples are taken in order to assess cotinine levels in plasma
Microcirculation assessment | 1 hour
  Microcirculation assessment is performed using the GlycoCheck system. This measures the endothelial cell surface layer non-invasively by applying a clinical videomicroscope to the sublingual arteries.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny A Bosson, MD;PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided